CLINICAL TRIAL: NCT00514813
Title: An Open-Label, Phase IV, Multi-Centre Study to Investigate the Long-Term Safety and Efficacy of Subcutaneous Dynepo in Adult Patients With Anaemia Associated With Chronic Kidney Disease
Brief Title: Dynepo Long-Term Safety Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The termination of the study is not linked to a product recall or result of any safety signal. Rather it was sponsor's commercial decision to withdraw the MA
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPD490-402; 2007-000054-31 (EudraCT Number)
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Anemia; Kidney Failure, Chronic
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — Erythropoietin; epoetin delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dynepo (Epoetin delta) (Experimental): Subjects received Dynepo (Epoetin delta) either twice weekly (BIW), once weekly (QW), once every 2 weeks (Q2W) or once every 4 weeks (Q4W) based on what is appropriate for the subject
  Interventions: Drug: Dynepo

INTERVENTIONS:
Drug: Dynepo — Subcutaneous injection either BIW, QW, Q2W or Q4W based on what is appropriate for the subject
  Other Names: Epoetin delta

SUMMARY:
To assess the incidence rate of Treatment Emergent Adverse Events (TEAEs) over 2 years in patients treated with Dynepo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who complete Dynepo study SPD490-301.
2. Patients who continue to require epoetin (EPO) treatment and have had a Hb level of 10g/dL between Weeks 16 and 24 of study SPD490-301.

Exclusion Criteria:

1. Withdrawal, before Week 24, from study SPD490-301.
2. Pregnant or lactating women.
3. Uncontrolled hypertension.
4. Thrombocytopenia (platelet count <75,000/mm3).
5. Active bleeding disorder (diathesis) (for example, gastrointestinal bleeding or genitourinary tract bleeding).
6. Treatment with immunosuppressive drugs (other than corticosteroids for a chronic condition) in the 30 days immediately prior to enrolment in this study.
7. Androgen therapy in the 30 days immediately prior to enrolment in this study.
8. Known Human Immunodeficiency Virus (HIV) infection.
9. History of hypersensitivity to Dynepo.
10. Known to have Ab against EPO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-06-06 (Actual); Primary Completion 2008-07-31 (Actual); Study Completion 2008-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Heilig Hartziekenhuis Department of Nephrology, Lier, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal.
Pre-assignment Details: Subjects received Dynepo (Epoetin delta) either twice weekly (BIW), once weekly (QW), once every 2 weeks (Q2W) or once every 4 weeks (Q4W) at a dose that is appropriate for them and not to exceed 20,000 IU at any one time.
Groups:
- Dynepo (Epoetin Delta) Twice Weekly (BIW): Epoetin delta (Dynepo) dosed twice-a-week
- Dynepo Once Weekly (QW): Epoetin delta dosed once-a-week
- Dynepo Once Every 2 Weeks (Q2W): Epoetin delta dosed once every 2 weeks
- Dynepo Once Every 4 Weeks (Q4W): Epoetin delta dosed once every 4 weeks
Period: Overall Study
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W)
Started | 15 | 86 | 47 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 86 | 47 | 4
Not completed — Study terminated | 14 | 74 | 40 | 2
Not completed — Adverse Event | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Kidney transplant | 0 | 6 | 2 | 0
Not completed — Death | 0 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W) | Total
Number analyzed (Participants) | 15 | 86 | 47 | 4 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 31 | 22 | 1 | 61
  >=65 years | 8 | 55 | 25 | 3 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.93) | 64.8 (13.7) | 65.2 (14.03) | 66.3 (21.39) | 64.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 33 | 16 | 2 | 58
  Male | 8 | 53 | 31 | 2 | 94
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 6 | 6 | 0 | 12
  Austria | 0 | 1 | 0 | 0 | 1
  France | 1 | 6 | 3 | 1 | 11
  Germany | 5 | 19 | 7 | 0 | 31
  Italy | 1 | 24 | 17 | 0 | 42
  Latvia | 3 | 7 | 3 | 0 | 13
  Spain | 0 | 8 | 8 | 3 | 19
  United Kingdom | 5 | 15 | 3 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Rate of Emergence of Treatment Emergent Adverse Events (TEAEs)
Time Frame: Over the course of 2 Years
Population: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal.
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Hemoglobin (Hb) Concentrations at 2 Years
Time Frame: Baseline and 2 years
Population: as for outcome 1
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Hematocrits at 2 Years
Time Frame: Baseline and 2 years
Population: as for outcome 1
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The adverse events were collected on the Safety Population defined as all subjects randomized who received at least one dose of Dynepo. Therefore, 150 of the 152 enrolled subjects constituted the Safety Population. Therefore, the second Arm has 84 subjects instead of 86 as shown in the participant flow.
Arm/Group | Dynepo (Epoetin Delta) Twice Weekly (BIW) | Dynepo Once Weekly (QW) | Dynepo Once Every 2 Weeks (Q2W) | Dynepo Once Every 4 Weeks (Q4W)
Serious Adverse Events (participants affected / at risk) | 1/15 | 14/84 | 6/47 | 1/4
Other Adverse Events (participants affected / at risk) | 7/15 | 62/84 | 32/47 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dynepo (Epoetin Delta) Twice Weekly (BIW) (N=15) | Dynepo Once Weekly (QW) (N=84) | Dynepo Once Every 2 Weeks (Q2W) (N=47) | Dynepo Once Every 4 Weeks (Q4W) (N=4)
Acute MI (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Catheter-related complication (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Dialysis device complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dynepo (Epoetin Delta) Twice Weekly (BIW) (N=15) | Dynepo Once Weekly (QW) (N=84) | Dynepo Once Every 2 Weeks (Q2W) (N=47) | Dynepo Once Every 4 Weeks (Q4W) (N=4)
Constipation (Gastrointestinal disorders) | 0 | 5 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 6 | 1
Nausea (Gastrointestinal disorders) | 0 | 5 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 6 | 2 | 0
Edema peripheral (General disorders) | 1 | 1 | 1 | 0
Vessel puncture site hematoma (General disorders) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 5 | 4 | 0
Nasopharyngitis (Infections and infestations) | 0 | 6 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0
Dialysis device complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hemaglobin decreased (Investigations) | 1 | 0 | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 6 | 2 | 1
Hypotension (Vascular disorders) | 0 | 3 | 3 | 1
Orthostatic hypertension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study terminated early due to a decision by Shire Pharmaceuticals to permanently cease marketing Dynepo due to commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.